CLINICAL TRIAL: NCT04007913
Title: Incorporating teleCBIT Into a Hospital-Based Tic Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Jose State University (Other)
Collaborators: American Academy of Neurology (Other); Tourette Association of America (Other)
Responsible Party: Principal Investigator, Matthew Capriotti, Assistant Professor, San Jose State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSCTRF2016
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Tic Disorders; Tourette Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Masking Description: True masking not possible due to single-arm design. However, independent evaluator is blind to treatment utilization and progress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- teleCBIT (Experimental): Patient receive eight sessions of individual teleCBIT, in accordance with Woods et al's (2008) protocol, from a licensed psychologist.
  Interventions: Behavioral: teleCBIT

INTERVENTIONS:
Behavioral: teleCBIT — Eight sessions of individual behavior therapy

SUMMARY:
This is a single-arm open trial of Comprehensive Behavioral Intervention for Tics (CBIT) delivered to pediatric and adult patients with persistent tic disorders in their homes via videoconferencing (i.e., teleCBIT). All participants who enroll will receive teleCBIT.

DETAILED DESCRIPTION:
Comprehensive Behavioral Intervention for Tics (CBIT) is a behavioral therapy with proven efficacy for treating persistent tic disorders (e.g., Tourette Syndrome) in youth and adults. Lack of access to a local CBIT provider prevents treatment access for many patients who could benefit from CBIT. Providing CBIT to patients in their homes via videoconferencing technology (i.e., teleCBIT) is a promising approach to increasing CBIT access. This study investigates treatment uptake, acceptability, feasibility, and clinical effectiveness of teleCBIT among pediatric and adult patients enrolled as patients in a state-of-the-art medical tic program.

ELIGIBILITY:
Inclusion Criteria:

* age 5-65, diagnosis of Tourette Syndrome or other persistent tic disorder (per diagnostic interview and self-report of prior physician diagnosis)
* Clinical Global Impressions - Severity Score > 3 (i.e., "moderately ill" or worse),
* unmedicated or on stable medication treatment for tics and psychiatric problems,
* fluency in English
* a functional accessible home computer and high speed (i.e., cable/DSL) internet connection
* willingness to sign a release of information to contact a local, licensed medical or mental health provider, of whom they are currently a patient (in case of emergent safety concerns).
* Minor participants must have a parent or guardian who is fluent in English available to attend treatment and assessment sessions.

Exclusion Criteria:

* significant suicidality, (i.e., a score of > 12 on the MINI or MINI-Kid suicidality module);
* prior diagnoses of intellectual disability; pervasive developmental disorder, mania, schizophrenia, psychotic disorder, substance abuse, substance dependence, or conduct disorder; currently experiencing a psychosocial, psychiatric, or neurological problem that requires immediate care
* lack of a functional home computer with high speed (i.e., cable or DSL) internet connection;
* or, prior receipt of >3 previous sessions of behavior therapy for tics within the past year (per self/parent report)

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Yale Global Tic Severity Scale Tic Severity Score (YGTSS) | Change from pre-treatment (i.e., week 0) to post-treatment (i.e., 10-week)
  YGTSS Tic Severity Score (0-50) as rated by independent evaluator. Higher scores indicate more severe tics.

SECONDARY OUTCOMES:
Clinical Global Impression: Improvement (CGI:I) Score | CGI:I score at post-treatment (Week 10), which assesses change from pre-treatment (i.e., week 0)
  CGI:I scores (range: 1-7) describe the global level of change in clinical severity of a disorder. Lower scores indicate more favorable change over time. Following common practice, we will also dichotomize CGI:I scores to evaluate Clinical Responder Status according to CGI:I score (i.e., responder: CGI:I=1 or 2; non-responder=CGI:I>2)
Parent Tic Questionnaire (PTQ) Total Tic Severity Score | Change from pre-treatment (i.e., week 0) to post-treatment (i.e., 10-week)
  Child Tic Severity as measured by parent-report on the PTQ (range: 0-224). Higher scores indicate more severe tics.
Adult Tic Questionnaire (ATQ) Total Tic Severity Score | Change from pre-treatment (i.e., week 0) to post-treatment (i.e., 10-week)
  Adult Tic Severity as measured by self-report on the ATQ (range: 0-224). Higher scores indicate more severe tics.
Yale Global Tic Severity Scale (YGTSS) Impairment Score | Change from pre-treatment (i.e., week 0) to post-treatment (i.e., 10-week)
  YGTSS Impairment Score (0-50) as rated by independent evaluator. Higher scores indicate greater tic-related impairment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Jose State University, San Jose, California
  - University of Florida Health, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Capriotti MR, Wellen BC, Young BN, Himle MB, Conelea CA, Espil FM, Simpson H, Mathews CA. Evaluating the feasibility, acceptability, and preliminary effectiveness of tele-comprehensive behavior therapy for tics (teleCBIT) for Tourette syndrome in youth and adults. J Telemed Telecare. 2025 Apr;31(3):328-337. doi: 10.1177/1357633X231189305. Epub 2023 Aug 7. PMID 37545359